CLINICAL TRIAL: NCT03996421
Title: Determination of Iron Absorption Mechanism From Ferrous Fumarate With Galacto-oligosaccharides Using Stable Isotope Appearance Curves
Brief Title: Determination of Iron Absorption Mechanism From Ferrous Fumarate With GOS
Acronym: Fe_GOS_3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Burgerstein Vitamine (Industry)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Principal Investigatior, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Fe_GOS_3
Record Dates: First submitted 2019-06-06; First posted 2019-06-24 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Low Iron Stores
Keywords: Low iron stores; Prebiotics; Galacto-oligosaccharides
MeSH Terms: interventions — ferrous fumarate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ferrous fumarate (Experimental): labelled iron as ferrous fumarate
  Interventions: Dietary Supplement: nutritional iron (14 mg) supplement in form of ferrous fumarate
- ferrous fumarate + 15 g GOS (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 15 g GOS
  Interventions: Dietary Supplement: ferrous fumarate + 15 g GOS

INTERVENTIONS:
Dietary Supplement: nutritional iron (14 mg) supplement in form of ferrous fumarate — nutritional iron (14 mg) supplement in form of ferrous fumarate
  Arms: ferrous fumarate
Dietary Supplement: ferrous fumarate + 15 g GOS — nutritional iron (14 mg) supplement in form of ferrous fumarate with addition of prebiotics (15 g GOS)
  Arms: ferrous fumarate + 15 g GOS

SUMMARY:
The aim is to investigate the mechanism by which galacto-oligosaccharide acutely increases iron absorption by using stable isotope appearance curves. This will allow the evaluation of changes in serum iron isotopes over the first few hours after administration of the iron supplement and provides information where and in what amount iron absorption takes place in the GI-tract.

DETAILED DESCRIPTION:
Iron is an important mineral in our body and fulfills essential functions such as for example oxygen transport from the lungs to the tissues. Iron deficiency is still the most common and widespread nutritional disorder in the world according to WHO. Common iron supplements all have their limitations in terms of availability and compatibility. Prebiotic fibers, such as galacto-oligosaccharides (GOS), selectively enhance growth of beneficial colonic bacteria. Prebiotics in general enhance the production of short-chain fatty acids (SCFAs) and thereby decrease luminal pH. Through the reduction in pH, prebiotics can enhance absorption of minerals such as calcium and magnesium and they have been proposed to potentially improve iron absorption.

In a recent iron absorption study in adult women with low iron stores in the laboratory of human nutrition ETH zurich, it was found that 15 g of GOS given with an iron supplement in the form of iron fumarate acutely increased iron absorption when given with water and a bread based meal. The dose of 15 g of GOS was tolerated well by the participants. As a follow up to the study, the aim of the current study is to investigate the mechanism by which GOS acutely increases iron absorption by using stable isotope appearance curves. This will allow the evaluation of changes in serum iron isotopes over the first few hours after administration of the iron supplement and provides information where and in what amount iron absorption takes place in the GI-tract.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* SF levels 15-30 µg/L
* Normal body Mass Index (18.5-24.9 kg/m2)
* Body weight <70 kg
* Signed informed consent

Exclusion Criteria:

* Severe anaemia (Hb < 80 g/L)
* Elevated CRP >10.0 mg/L
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole studies (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration, including pre- and-or probiotics supplements (excluding foods and beverages with life cultures such as yoghurt, raw milk cheese and kombucha)
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Difficulties with blood sampling
* Use of antibiotics over the past month
* Known hypersensitivity to iron supplements in the given amount, GOS, or lactose
* Women who are pregnant or breast feeding
* Women who intend become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, inject-able, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse -
* Smokers (> 1 cigarette per week)
* Inability to follow the procedures of the study, e.g. due to language problems, self-- reported psychological disorders, etc. of the participant
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are being studied
Enrollment: 12 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
serum iron isotope concentration | 29 days
  serum iron isotope concentration from ferrous fumarate with or without the addition of GOS at all the different time points. Serum iron isotope concentration absorbed from the iron supplements will be calculated based on the shift of the iron isotope ratios in the collected blood samples at least 14 days after the last administration of the isotopically labelled supplements.The iron isotope ratios in the collected blood samples will be measured using an ICP-mass spectrometry instrument (NEPTUNE, Thermo Finnigan).
total fractional iron absorption | 29 days
  total iron fractional absorption from ferrous fumarate with or without the addition of GOS at all the different time points. Fractional absorption of iron (%) from the iron supplements will be calculated based on the shift of the iron isotope ratios in the collected blood samples at least 14 days after the last administration of the isotopically labelled supplements.The iron isotope ratios in the collected blood samples will be measured using an ICP-mass spectrometry instrument (NEPTUNE, Thermo Finnigan).

SECONDARY OUTCOMES:
Haemoglobin (Hb) | 29 days
  Haemoglobin (Hb) (g/L)
serum ferritin (SF) | 29 days
  serum ferritin (SF) (microg/L)
serum transferrin receptor (sTfR) | 29 days
  serum transferrin receptor (sTfR) (mg)L)
alpha-1-acid glycoprotein (AGP) | 29 days
  alpha-1-acid glycoprotein (AGP) (g/L)
C - reactive protein (CRP) | 29 days
  C - reactive protein (CRP) (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, Dr., Principal Investigator — Laboratory of Human Nutrition ETH Zürich
Locations (1):
- Laboratory of Human Nutrition, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeroense FMD, Michel L, Zeder C, Herter-Aeberli I, Zimmermann MB. Consumption of Galacto-Oligosaccharides Increases Iron Absorption from Ferrous Fumarate: A Stable Iron Isotope Study in Iron-Depleted Young Women. J Nutr. 2019 May 1;149(5):738-746. doi: 10.1093/jn/nxy327. PMID 31004135
- [Derived] Husmann FMD, Stierli L, Bram DS, Zeder C, Kramer SD, Zimmermann MB, Herter-Aeberli I. Kinetics of iron absorption from ferrous fumarate with and without galacto-oligosaccharides determined from stable isotope appearance curves in women. Am J Clin Nutr. 2022 Mar 4;115(3):949-957. doi: 10.1093/ajcn/nqab361. PMID 34726703